CLINICAL TRIAL: NCT04147494
Title: PET Biodistribution Study of 68Ga-PSMA-11 and 68Ga-FAPI-46 in Patients With Non-Prostate Cancers: An Exploratory Biodistribution Study With Histopathology Validation
Brief Title: Experimental PET Imaging Scans Before Cancer Surgery to Study the Amount of PET Tracer Accumulated in Normal and Cancer Tissues
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Society of Nuclear Medecine and Molecular Imaging (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-000756; NCI-2019-07265 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-10-24; First posted 2019-11-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma; Colon Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Head and Neck Carcinoma; Kidney Carcinoma; Lung Carcinoma; Ovarian Carcinoma; Pancreatic Carcinoma; Solid Neoplasm; Uterine Corpus Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms | interventions — FAPI-46; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Basic Science (68Ga-FAPi-46 PET/CT, 68Ga-PSMA-11 PET/CT) (Experimental): Patients receive 68Ga-FAPi-46 intravenously (IV), and then undergo PET/computed tomography (CT) over 20-90 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable). Patients may also receive 68Ga-PSMA-11 IV and undergo PET/CT scan over 20-50 minutes on a separate day (for volunteer patients only, PSMA PET/CT is optional and not required).
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga 68 FAPi-46; Radiation: Gallium Ga 68-labeled PSMA-11; Procedure: Positron Emission Tomography; Radiation: 18F-FDG

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT scan; tomography
Radiation: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: 68Ga-FAPi-46; Gallium-68-FAPi-46
Radiation: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: 18F-FDG — Given IV
  Other Names: 18F-fluorodeoxyglucose

SUMMARY:
This phase I trial studies a new imaging technique called FAPi PET/CT to determine where and to which degree the FAPI tracer (68Ga-FAPi-46) accumulate in normal and cancer tissues in patients with non-prostate cancer. The research team also want to know whether what they see on PET/CT images represents the tumor tissue being excised from the patient's body. The research team is also interested to investigate another new imaging technique called PSMA PET/CT. Participants will be invited to undergo another PET/CT scan, with the PSMA tracer (68Ga-PSMA-11). This is not required but just an option for volunteer patients. Patients who have not received an 18F-FDG PET/CT within one month of enrollment will also undergo an FDG PET/CT scan. The PET/CT scanner combines the PET and the CT scanners into a single device. This device combines the anatomic (body structure) information provided by the CT scan with the metabolic information obtained from the PET scan. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of, in the case of this research, 68Ga-PSMA-11 and 68Ga-FAPi, and 18F-FDG (if applicable). Because some cancers take up 68Ga-PSMA-11 and/or 68Ga-FAPi it can be seen with PET. CT utilizes x-rays that traverse the body from the outside. CT images provide an exact outline of organs where it occurs in patient's body. FAP stands for Fibroblast Activation Protein. FAP is produced by cells that surround tumors. The function of FAP is not well understood but imaging studies have shown that FAP can be detected with FAPI PET/CT. Imaging FAP with FAPI PET/CT may in the future provide additional information about various cancers. PSMA stands for Prostate Specific Membrane Antigen. This name is incorrect as PSMA is also found in many other cancers. The function of PSMA is not well understood but imaging studies have shown that PSMA can be detected with PET in many non-prostate cancers. Imaging FAP with PET/CT may in the future provide additional information about various cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of gallium Ga 68 FAPi-46 (68Ga-FAPi-46) and gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) in normal and cancer tissues of patients with various non-prostate malignancies. The goal is to determine where and to which degree 68Ga-FAPi-46 and 68Ga-PSMA-11 accumulates in normal and cancer tissues.

SECONDARY OBJECTIVES:

I. To evaluate whether 68Ga-FAPi-46 and 68Ga-PSMA-11 accumulation observed by positron emission tomography (PET) correlates with the amount of fibroblast activation protein (FAP) and prostate specific membrane antigen (PSMA) in excised cancer tissue, respectively.

II. To evaluate the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution (when available) to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-).

EXPERIMENTAL OBJECTIVE:

III. Assess the 68Ga-FAPI-46 biodistribution correlation with 68Ga-PSMA-11, if the patient volunteers for optional scan, and 18F-fluodeoxyglucose (FDG), if any FDG PET/computed tomography (CT) has been performed as standard-of-care.

OUTLINE:

Patients receive 68Ga-FAPi-46 intravenously (IV) and undergo PET/CT scan over 20-50 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable). Patients may also receive 68Ga-PSMA-11 IV and undergo PET/CT scan over 20-50 minutes on a separate day (for volunteer patients only, PSMA PET/CT is optional and not required).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following cancer types:

  * Breast cancer
  * Colon cancer
  * Esophageal cancer
  * Gastric cancer
  * Head and Neck cancer
  * Lung cancer
  * Ovarian cancer
  * Pancreatic cancer
  * Renal cancer
  * Uterus cancer
* Patients who are scheduled to undergo surgical resection of the primary tumor and/or metastasis
* Patient can provide written informed consent
* Patient is capable of complying with study procedures
* Patient is able to remain still for duration of imaging procedure (up to one hour)

Exclusion Criteria:

* Patient is pregnant or nursing
* Patients with any new cancer therapy between the baseline 18F-FDG PET/CT and the investigational FAPI PET/CT
* Patient has underlying disease which, based on the judgment of the investigator, might interfere with the collection of high quality data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-10-17 (Estimated)

PRIMARY OUTCOMES:
To define and document the biodistribution of gallium Ga 68 FAPi-46 (68Ga-FAPi-46) and gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) in normal and cancer tissues of patients with various non-prostate malignancies | 60 minutes after tracer injection
  To quantify tumor tissue and normal background organs positron emission tomography (PET) tracer uptake by semi-quantitative analysis (unit/metrics = standardized uptake values (SUV)). The 68Ga-PSMA-11 and 68Ga-FAPI-46 tracer biodistribution will be described by mean and maximum standardized uptake values (SUVmean and SUVmax).

SECONDARY OUTCOMES:
68Ga-FAPi-46 and 68Ga-PSMA-11 accumulation | From date of imaging to date of surgery (range 1-60 days)
  To evaluate whether 68Ga-FAPi-46 accumulation observed by PET correlates with the amount of FAP in excised cancer tissue as assessed by immunohistochemistry (IHC).
evaluate the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution | up to 2 years
  2. To evaluate the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution (when available) to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-).

OTHER OUTCOMES:
Additional correlation of biodistribution of standard of care tracer | 60 minutes after tracer injection
  assess the 68Ga-FAPI-46 biodistribution correlation with 68Ga-PSMA-11, if the patient volunteers for optional scan

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- Ethan Lam, Los Angeles, California, United States

REFERENCES:
- [Derived] Kunikowska J, Bizon M, Pelka K, Derlatka P, Olszewski M, Krolicki L. 68 Ga-Prostate-Specific Membrane Antigen PET/CT in Ovarian Tumors : Potential to Differentiate Benign and Malignant Tumors Before Surgery: A Preliminary Report. Clin Nucl Med. 2023 Feb 1;48(2):e60-e66. doi: 10.1097/RLU.0000000000004486. Epub 2022 Nov 18. PMID 36512649